CLINICAL TRIAL: NCT06871098
Title: Evaluating the Founder Exercise Technique: Improving Mechanics and Confidence in the Hip Hinge
Brief Title: Improving Mechanics and Confidence in the Hip Hinge
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Florida (Other)
Responsible Party: Principal Investigator, William J. Hanney, Professor, University of Central Florida
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00007247
Record Dates: First submitted 2025-02-13; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-02

CONDITIONS: Hip Hinge; Hip and Knee Movement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hip Hinge (Experimental): * Each participant will receive 8 minutes of instruction from Assessor 2 on performing the Founder Exercise according to the standardized training strategies documented in the attached file labeled "Founder Exercise Instruction".
  * The participant will then be allowed 10 practice repetitions with cueing from Assessor 2. Guidelines for cuing can be found in the "Founder Exercise Instruction" document.
  Interventions: Other: Hip Hinge Instruction

INTERVENTIONS:
Other: Hip Hinge Instruction — The participant will be instructed to perform a hip hinge movement based on their current understanding and ability. This initial movement assessment will serve as a baseline measure to analyze the participant's natural hip hinge mechanics before any intervention. The purpose of this assessment is to determine whether the implementation of the Founder Exercise intervention leads to significant changes in the kinematics of the hip hinge movement.

SUMMARY:
To evaluate if the Founder exercise will significantly change participants kinematics when performing hip hinge movement. Secondary purpose is to evaluate if completing the Founder Exercise intervention will improve confidence in performing a hip hinge.

DETAILED DESCRIPTION:
Procedures Involved*

* This study will employ a Single Group Pre-Post Test Design. Baseline data will be collected from all participants prior to the intervention. Participants will then undergo the intervention, after which the same measures will be administered to evaluate changes attributable to the intervention.
* The intervention will be administered in one session to each participant individually by a team of UCF DPT students (Assessor 1 and 2) in person at University of Central Florida's Health & Science Building I Room 231. Each session will be divided into 3 phases: (I) Pre-intervention assessment, (II) Intervention, (III) Post-intervention assessment.

Pretest:

1. The participant will be asked to provide their age, biological sex, self-reported height, and self-reported weight. The participant will be assigned a subject ID number (These will be sequential, starting at P001).
2. The participant will be asked to fill out a paper copy of a patient confidence scale (attached document labeled "Patient Confidence Scale") for utilizing a hip hinge movement pattern. The scale will consist of Likert-type questions, asking participants to rate their confidence in performing the hip hinge during a range of functional tasks, such as lifting, bending, and squatting. Each question will be rated on a 5-point scale, with higher scores indicating greater confidence in safely executing the movement.
3. Participants will be asked to remove their socks and shoes to allow for the precise placement of reflective markers (small skin-safe adhesive stickers). A trained member of the research team will position these markers either directly on the skin or over clothing at specific anatomical landmarks on the left side of the body. The landmarks include: the lateral epicondyle of the humerus, the head of the humerus, the greater trochanter, the lateral joint line of the knee, and the lateral malleolus
4. The participant will then be instructed using the following statement: "Please perform a hip hinge movement based on your current understanding and ability". Assessor 1 will obtain the following measurements:

   Foot placement: The participant will step on to the prepared surface (a sheet of paper that has been rolled out and secured to the ground with tape). The participant will stand with both feet on the paper and instructed to adjust to their preferred start position as necessary. Assessor 1 will mark the paper at the center of each calcanei and at the distal end of each great toe. At the conclusion of the movement the participant will step off the paper and Assessor 1 will measure the distance between the two center points using a tape measure to obtain the participant's stance width. Assessor 1 will then use a goniometer to measure the angle between the center point and the great toe point of each foot to obtain the angle of orientation of the foot.

   Shoulder flexion, hip flexion, knee flexion, ankle sagittal plane flexion: The angles will be measured using 2D video analysis through the OnForm app on an iPad. This will be recorded directly into the app and stored by OnForm (OnForm's privacy policy is attached). This app enables video recording and allows for detailed frame-by-frame analysis, including precise marking of anatomical structures and the calculation of distances and angles during the participant's hip hinge movement. The iPad will be positioned to the left of the participant so that all reflective markers are in view of the camera when the arms are raised overhead.

   o Then, the participant's grip strength will be measured using a hand grip dynamometer, a reliable and valid tool for measuring isometric grip force. The participant will stand with the test arm bent at the elbow to 90 degrees with the forearm and wrist in neutral. The dynamometer will be placed in the test hand and the participant will be instructed to perform a maximal squeeze. This will be repeated 3 times, and the highest measure will be documented. This will then be repeated for the opposite hand.

   Intervention:

   o Each participant will receive 8 minutes of instruction from Assessor 2 on performing the Founder Exercise according to the standardized training strategies documented in the attached file labeled "Founder Exercise Instruction".

   o The participant will then be allowed 10 practice repetitions with cueing from Assessor 2. Guidelines for cuing can be found in the "Founder Exercise Instruction" document.

   Post Test:

   o The participant will perform a final hip hinge during which all measurements will be obtained by Assessor 1 identically as in the pre-test.
   * Grip strength will be reassessed.
   * The participant will be asked to complete a new paper copy of the patient confidence scale.
   * In order to lessen the probability or magnitude of risks, all participants will be screened for low back pain, pelvic pain, and hip pain prior to administration of the intervention. This will be accomplished by a member of the research team verbally asking the following question: "Are you currently experiencing any low back pain, pelvic pain, and/or hip pain?" Participants will also be supervised by the assessors throughout the intervention to ensure safety.

   Sharing of Results with Subjects*

   • Individual subject results will only be shared with participants by request at the completion of the study. They will receive access to their data electronically via email.

   Study Timelines*
   * Participants will conclude their participation in one 45 minute session. They will complete the pretest measurements, intervention, and posttest measurements within this window of time.
   * The goal of this study is to complete enrollment by the end of the Summer, 2025 semester.
   * The estimated date for investigators to complete primary analyses is by the end of the Fall, 2025 semester.

   Inclusion and Exclusion Criteria*

   • Participants will be screened for eligibility by responding to an email sent by the research team. (This email is attached and labeled as "Participant Eligibility Confirmation Email").
   * Inclusion Criteria:

     o Age between 18 and 50 years.

     o Ability to perform physical exercises, including bending at the waist.
     * Ability to understand verbal and tactile cues.
   * Exclusion Criteria:

     o History of low back pain, pelvic pain, or hip pain.

     o Participants that have pain with the intervention.

     o Current or past musculoskeletal injuries affecting hip, knee, ankle, or foot function.
     * Any condition limiting the ability to perform or participate in physical activities.
     * Pregnant individuals or those planning pregnancy during the study duration.
     * This project will exclude the following special populations from participating: Adults unable to consent, individuals who are not yet adults (infants, children, teenagers), pregnant women, and prisoners. Pregnant women will be excluded due to the natural change in body mechanics that occurs during pregnancy, as this would lead to outliers in the data.

   Local Number of Subjects • A total number of 30 participants will be needed to complete this study, however, we will enroll 33 in order to account for an anticipated 10% attrition rate.

   Recruitment Methods
   * Recruitment will begin immediately after IRB approval.
   * Participants will be recruited from the general population of the greater UCF community. This will include students, faculty and staff.
   * Subjects will be recruited via physical and virtual flyers. Physical flyers will be posted on campus or distributed by hand in classrooms. Virtual flyers will be shared by email and social media via postings on Instagram from the professional UCF DPT account. The flyer is located in an attached document ("Hip Hinge Flyer 3").
   * Digital advertisement on the College of Health Professions and Sciences Research Participant Website. (Same as the uploaded flyer). (https://healthprofessions.ucf.edu/research/studies/)
   * Once individuals express interest in taking part in the study, they will be contacted via email by the investigators to confirm eligibility using the inclusion/exclusion criteria (see the document labeled "Participant Eligibility Confirmation Email").
   * Compensation will not be provided to subjects as part of this study.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 50 years.
* Ability to perform physical exercises, including bending at the waist.
* Ability to understand verbal and tactile cues.

Exclusion Criteria:

* History of low back pain, pelvic pain, or hip pain.
* Participants that have pain with the intervention.
* Current or past musculoskeletal injuries affecting hip, knee, ankle, or foot function.
* Any condition limiting the ability to perform or participate in physical activities.
* Pregnant individuals or those planning pregnancy during the study duration.
* This project will exclude the following special populations from participating: Adults unable to consent, individuals who are not yet adults (infants, children, teenagers), pregnant women, and prisoners. Pregnant women will be excluded due to the natural change in body mechanics that occurs during pregnancy, as this would lead to outliers in the data.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-03 (Estimated); Primary Completion 2025-08-25 (Estimated); Study Completion 2026-03-23 (Estimated)

PRIMARY OUTCOMES:
2D motion capture | immediately after the intervention/procedure
  The angles will be measured using 2D video analysis through the OnForm app on an iPad. This will be recorded directly into the app and stored by OnForm (OnForm's privacy policy is attached). This app enables video recording and allows for detailed frame-by-frame analysis, including precise marking of anatomical structures and the calculation of distances and angles during the participant's hip hinge movement. The iPad will be positioned to the left of the participant so that all reflective markers are in view of the camera when the arms are raised overhead.
Grip Strength | immediately after the intervention/procedure
  the participant's grip strength will be measured using a hand grip dynamometer, a reliable and valid tool for measuring isometric grip force. The participant will stand with the test arm bent at the elbow to 90 degrees with the forearm and wrist in neutral. The dynamometer will be placed in the test hand and the participant will be instructed to perform a maximal squeeze. This will be repeated 3 times, and the highest measure will be documented. This will then be repeated for the opposite hand.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Central Florida, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided